CLINICAL TRIAL: NCT03945695
Title: Pneumatic Vitreolysis Using the Drinking Bird Technique for Management of Vitreomacular Traction. A Prospective, Non-randomized, Interventional Study.
Brief Title: Pneumovitreolysis for Vitreomacular Traction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of location, unsatisfactory preliminary results
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Martin Kowalski, Principal investigator, University of Split, School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2181-147-01/06/M.S.-19-2
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2019-05

CONDITIONS: Vitreomacular Traction Syndrome
Keywords: VMT; VMA; Vitreomacular Adhesion; Pneumatic Vitreolysis

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, non-blinded, interventional single-arm pilot study.
Masking Description: non-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pneumatic Vitreolysis (Experimental): All included eyes will receive one intravitreal injection of filtered sulfur hexafluoride gas (SF6).
  Interventions: Procedure: Pneumatic Vitreolysis in combination with "Drinking-Bird-Technique"

INTERVENTIONS:
Procedure: Pneumatic Vitreolysis in combination with "Drinking-Bird-Technique" — 1. Appropriate anesthesia and antiseptic preparation of the surgical field
  2. Prophylactic paracentesis of the anterior chamber
  3. One intravitreal injection of 0.2 to 0.3 ml of filtered sulfur hexafluoride gas (SF6) into the test eye Remark: Intraocular pressure of the examined eye is to be controlled before the intervention and kept at an appropriate level after paracentesis by manual application of pressure.
  4. Patients are instructed to avoid supine position and to lie on one side or the abdomen during sleep until complete resorption of intraocular gas occured. In this period they should bend over several times during the day up to an angle of 90º or as much as possible, resembling the movement of a bird drinking water. (Hence the name "drinking-bird-technique".)
  Other Names: Pneumovitreolysis

SUMMARY:
In this prospective, non-randomized, single-arm pilot study, conducted at the Eye Clinic of the University Hospital Split, the investigators are going to evaluate the utility of a single intravitreal injection of sulfur hexafluoride in the treatment of patients with symptomatic vitreomacular traction. Following the injection patients are going to be instructed to bend forward several times a day, resembling a drinking bird, hence the name of this maneuver. The investigators plan to include approximately ten eyes, which will be followed up for a three month period. Outcome measures will be common parameters, like adhesion resolution, also to increase comparability with previously conducted studies. The collected data will be used to get an impression of the efficacy and safety of this intervention. Furthermore it will aid in the performance of a power analysis to determine an appropriate sample size for later larger studies.

DETAILED DESCRIPTION:
The Ethical Committee of the Split Clinical Hospital Center previously already gave consent for the conduction of this research. Any personal data obtained in this research was and will be kept and handled strictly confidential and according to the Medical Code of Ethics. All reports generated on the basis of this study will utilize the data of a sample of patients with the diagnosis of vitreomacular traction fulfilling the eligibility criteria prior to intervention. The purpose of the examinations, procedures, possible advantages, disadvantages and possible side effects of the intervention will be explained to all participants, possible questions are going to be answered and a signed informed consent obtained.

Patients are going to be selected by the study chair from his pool of patients according to the criteria of inclusion and exclusion, as stated below. After obtaining informed consent all patients will be assigned into the intervention group and receive treatment according to our predefined procedural protocol. Neither participants nor researchers will be blinded during the whole course of the study.

One of the investigators carries out regular control examinations at one week after the procedure, and then every 2 to 4 weeks thereafter. During each control examination visual acuity and intraocular pressure will be measured, moreover biomicroscopy, indirect ophthalmoscopy, and macular OCT (Cirrus OCT 5000 HD, Zeiss) of the treated eye are going to be performed. The following data are also going to be recorded by the same investigator: patient demographics (age, gender, right eye in relation to left eye), period of intravitreal injection of gas to the separation of the posterior vitreous body (PVD) and monitoring time. Any adverse events that have occurred after gas injection, including eye complications (eg. retinal tear or ablation, infections, increase in intraocular pressure, uveitis, bleeding and damage to the optic nerve), and systemic complications, are going to be recorded.

Statistical Analysis will be performed using IBM SPSS©. Descriptive Statistics will include patient demographic data and baseline characteristics. The mean, standard deviations, median, minimum, and maximum will be reported for continuous variables, whereas frequencies and proportions are going to be described for categorical variables. The investigators will furthermore utilize the collected data to perform a power analysis and determine an appropriate sample size for future studies evaluating the utility of a single intravitreal injection of SF6 in the management of symptomatic vitreomacular traction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* able to give written informed consent to the procedure
* diagnosis of symptomatic VMT based on clinical and OCT-findings

Exclusion Criteria:

* any form of retinal tear, macular degeneration, vascular occlusion of the retina, aphakia, high myopia (> -8 diopters), uncontrolled glaucoma, vitreous opacities, retinal ablation, previous vitrectomy surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Resolution of VMT | Three months
  Primary outcome measure is going to be resolution of vitreomacular traction as determined by OCT.

SECONDARY OUTCOMES:
Best corrected visual acuity improvement | One week, two weeks, one month, three months
  Visual acuity is going to be measured preoperatively, as well as on each control visit one week, two weeks, one month and three months post-intervention using standard testing by Snellen-chart.
Foveal outline | One week, two weeks, one month, three months
  Foveal outline is going to be described preoperatively, as well as on each control visit one week, two weeks, one month and three months post-intervention using OCT.
Central foveal thickness | One week, two weeks, one month, three months
  Central foveal thickness is going to be measured preoperatively, as well as on each control visit one week, two weeks, one month and three months post-intervention using OCT.
Maximum central foveal thickness | Three months
  Maximum central foveal thickness during the three-month follow-up period is going to be determined using regular OCT measurements.
Time needed for resolution | Three months
  Individual and average time needed for resolution of VMT after intervention will be described.
Side-effects | Three months
  All side-effects will be noted during the three-month follow-up period. Patients will be informed before intervention about possible side-effects and asked on every control-visit about occurrence.
Occurrence of retinal tear or ablatio | Three months
  Any occurrence of retinal tear or ablatio will be checked for utilizing OCT, included in our report and treated appropriately.
Number of patients recommended to undergo further therapy by vitrectomy | Three months
  In the case vitrectomy surgery seems to be necessary for further management, patients will be informed and recommended to continue further operative treatment. The number of patients referred to surgery will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ljubo Znaor, Assist. Prof., MD, PhD, Principal Investigator — Department of Ophthalmology, University Hospital of Split
Locations (1):
- University Hospital of Split, Department of Ophthalmology, Split, Croatia

IPD SHARING:
Plan to Share IPD: No
We are not going to share any personal participant data. Individual participant data will be anonymously included in the statistical analysis and reported accordingly.

REFERENCES:
- [Background] Chang LK, Fine HF, Spaide RF, Koizumi H, Grossniklaus HE. Ultrastructural correlation of spectral-domain optical coherence tomographic findings in vitreomacular traction syndrome. Am J Ophthalmol. 2008 Jul;146(1):121-7. doi: 10.1016/j.ajo.2008.03.001. Epub 2008 Apr 25. PMID 18439563
- [Background] Steel DH, Downey L, Greiner K, Heimann H, Jackson TL, Koshy Z, Laidlaw DA, Wickham L, Yang Y. The design and validation of an optical coherence tomography-based classification system for focal vitreomacular traction. Eye (Lond). 2016 Feb;30(2):314-24; quiz 325. doi: 10.1038/eye.2015.262. Epub 2016 Jan 15. PMID 26768921
- [Background] Duker JS, Kaiser PK, Binder S, de Smet MD, Gaudric A, Reichel E, Sadda SR, Sebag J, Spaide RF, Stalmans P. The International Vitreomacular Traction Study Group classification of vitreomacular adhesion, traction, and macular hole. Ophthalmology. 2013 Dec;120(12):2611-2619. doi: 10.1016/j.ophtha.2013.07.042. Epub 2013 Sep 17. PMID 24053995
- [Background] Stalmans P, Duker JS, Kaiser PK, Heier JS, Dugel PU, Gandorfer A, Sebag J, Haller JA. Oct-based interpretation of the vitreomacular interface and indications for pharmacologic vitreolysis. Retina. 2013 Nov-Dec;33(10):2003-11. doi: 10.1097/IAE.0b013e3182993ef8. PMID 23881226
- [Background] Bottos JM, Elizalde J, Rodrigues EB, Maia M. Current concepts in vitreomacular traction syndrome. Curr Opin Ophthalmol. 2012 May;23(3):195-201. doi: 10.1097/ICU.0b013e328352404c. PMID 22450220
- [Background] Folk JC, Adelman RA, Flaxel CJ, Hyman L, Pulido JS, Olsen TW. Idiopathic Epiretinal Membrane and Vitreomacular Traction Preferred Practice Pattern((R)) Guidelines. Ophthalmology. 2016 Jan;123(1):P152-81. doi: 10.1016/j.ophtha.2015.10.048. Epub 2015 Nov 12. PMID 26578445
- [Background] Dimopoulos S, Bartz-Schmidt KU, Gelisken F, Januschowski K, Ziemssen F. Rate and timing of spontaneous resolution in a vitreomacular traction group: should the role of watchful waiting be re-evaluated as an alternative to ocriplasmin therapy? Br J Ophthalmol. 2015 Mar;99(3):350-3. doi: 10.1136/bjophthalmol-2014-304961. Epub 2014 Oct 23. PMID 25342274
- [Background] Neffendorf JE, Simpson ARH, Steel DHW, Desai R, McHugh DA, Pringle E, Jackson TL. Intravitreal gas for symptomatic vitreomacular adhesion: a synthesis of the literature. Acta Ophthalmol. 2018 Nov;96(7):685-691. doi: 10.1111/aos.13547. Epub 2017 Aug 31. PMID 28857483
- [Background] Ochoa-Contreras D, Delsol-Coronado L, Buitrago ME, Velasco-Barona C, Quiroz-Mercado H. Induced posterior vitreous detachment by intravitreal sulfur hexafluoride (SF6) injection in patients with nonproliferative diabetic retinopathy. Acta Ophthalmol Scand. 2000 Dec;78(6):687-8. doi: 10.1034/j.1600-0420.2000.078006687.x. PMID 11167234
- [Background] Rodrigues IA, Stangos AN, McHugh DA, Jackson TL. Intravitreal injection of expansile perfluoropropane (c(3)f(8)) for the treatment of vitreomacular traction. Am J Ophthalmol. 2013 Feb;155(2):270-276.e2. doi: 10.1016/j.ajo.2012.08.018. Epub 2012 Nov 17. PMID 23164159
- [Background] Jorge R, Costa RA, Cardillo JA, Uno F, Bonomo PP, Farah ME. Optical coherence tomography evaluation of idiopathic macular hole treatment by gas-assisted posterior vitreous detachment. Am J Ophthalmol. 2006 Nov;142(5):869-71. doi: 10.1016/j.ajo.2006.05.062. PMID 17056375
- [Background] Steinle NC, Dhoot DS, Quezada Ruiz C, Castellarin AA, Pieramici DJ, See RF, Couvillion SC, Nasir MA, Avery RL. TREATMENT OF VITREOMACULAR TRACTION WITH INTRAVITREAL PERFLUOROPROPANE (C3F8) INJECTION. Retina. 2017 Apr;37(4):643-650. doi: 10.1097/IAE.0000000000001237. PMID 27681001
- [Background] Chan CK, Crosson JN, Mein CE, Daher N. PNEUMATIC VITREOLYSIS FOR RELIEF OF VITREOMACULAR TRACTION. Retina. 2017 Oct;37(10):1820-1831. doi: 10.1097/IAE.0000000000001448. PMID 28099316